CLINICAL TRIAL: NCT07376681
Title: Fertility Outcomes In Young Breast Cancer Patients And Their Prognosis And Offspring Health
Status: Enrolling by invitation | Type: Observational
Sponsor: Taizhou Hospital (Other)
Collaborators: Second Affiliated Hospital, Sun Yat-Sen University (Other); Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhang Yuzhu, attending doctor, Taizhou Hospital
Other Study IDs: ZYuzhu
Record Dates: First submitted 2025-11-26; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Prognosis; Fertility; Breast Cancer; Young People
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to clarify the fertility status of young breast cancer patients, verify the independent impact of fertility behavior on the prognosis of patients with different molecular types, and evaluate the association between treatment regimens and offspring health.

DETAILED DESCRIPTION:
This was a multicenter retrospective study on fertility outcomes and their prognosis and offspring health in young breast cancer patients. Based on the breast cancer database, the investigators registered the baseline data of young breast cancer patients (≤40 years old), including age at initial diagnosis, molecular typing, tumor stage, treatment plan, fertility protection measures, etc., and followed up by telephone/email and other means to collect their fertility status, recurrence and offspring growth and development data. The primary endpoints were the disease-free survival (DFS), overall survival (OS) after childbirth and childrens' growth and development. The secondary endpoints were the patient's fertility live birth rate, pregnancy outcomes and complications, use of fertility preservation techniques, breastfeeding status, etc. The investigators used the Kaplan-Meier method to draw the survival curve of the patients after childbirth, and analyzed the growth trajectory of the offspring born after diagnosis by the Lambda-Mu-Sigma method, and plotted the growth and development curve.The investigators used Log-rank to test the significance of differences in pregnancy rates between variables. The investigators used Univariate Cox regression analysis to screen factors related to prognosis, and then used multivariate Cox regression analysis to adjust for potential confounding factors to clarify independent prognostic indicators of disease. Finally, descriptive analyses were performed for other secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

Only subjects who meet all of the following inclusion criteria can be enrolled in this trial:

1. Female patients diagnosed with breast cancer aged ≤ 40 years;
2. Patients with pathologically confirmed breast cancer, and TNM stage 0-III, the disease is in a stable or progressive state;
3. Complete medical records and clinical follow-up data were available. Informed consent.

Exclusion Criteria:

Anyone who has one of the following conditions cannot be included in this trial:

1. Female patients with a diagnosis age>40 years;
2. Stage IV breast cancer at first diagnosis;
3. The presence of other reproductive system diseases caused by oligomenorrhea or amenorrhea and infertility; Loss of clinical data or loss to follow-up.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young breast cancer (≤40years)
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The overall-surviva(OS) period of childbirth after diagnosis | About 2 years after the start of the research.
  The starting time of OS regarded as after completing the childbearing behavior.Death is regarded as the end time of OS.
The disease-free survival(DFS) period of childbirth after diagnosis | About 2 years after the start of the research
  The starting time of DFS is regarded as after completing the childbearing behavior.Repase or distant metastasis is regarded as the end time of DFS.
The growth and development of offspring | About 2 years after the start of the research
  The growth and development of young breast cancer patients after diagnosis. By collecting their height, weight and other data, using the Lambda-Mu-Sigma method recommended by WHO, the obtained data is fitted to the offspring growth curve of young breast cancer patients and compared with the standard curve, in order to evaluate whether the patients' offspring grows abnormally.
The occurrence of diseases in the descendants of young breast cancer patients. | About 2 years after the start of the research
  Descriptive research. Describe the number of serious disease events in the offspring of young breast cancer patients after diagnosis, such as the number of secondary tumors in childhood

SECONDARY OUTCOMES:
Fertility rate of young breast cancer patients. | About 2 years after the start of the research.
  The ratio of the number of young breast cancer patients giving birth after diagnosis to the total number of samples included.
Complications during pregnancy after diagnosis of young breast cancer patients. | About 2 years after the start of the research
  Descriptive research. Describe the complications during pregnancy after the diagnosis of young breast cancer patients, and describe the specific types and proportion of complications.
The use of fertility preservation in the reproductive process of young breast cancer patients. | About 2 years after the start of the research
  Descriptive research. Count the proportion of young breast cancer patients who use fertility preservation technology during pregnancy after diagnosis.
Breastfeeding. | About 2 years after the start of the research.
  It mainly describes the proportion of patients breastfeeding and whether there are any difficulties due to the disease in the process.

CONTACTS AND LOCATIONS:
Overall Officials: Yuzhu Zhang, Principal Investigator — Taizhou Hospital
Locations (1):
- Taizhou Central Hosipital, Taizhou, Zhejiang, China